CLINICAL TRIAL: NCT02364882
Title: A Phase 1, Open-Label, Within-Subject Dose-Escalation Study to Evaluate the Clinical Vulvar-Vaginal Safety and Pharmacokinetic Profile of SST-6006, a Topical Sildenafil Cream (5% w/w), in Healthy Postmenopausal Women
Brief Title: A Open-Label, Within-Subject Dose-Escalation Study to Evaluate the Clinical Safety and Pharmacokinetic Profile of a Topical Sildenafil Cream (5% w/w), in Healthy Postmenopausal Women
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Strategic Science & Technologies, LLC (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None
Other Study IDs: SST-6006-008-01
Record Dates: First submitted 2015-01-27; First posted 2015-02-18 (Estimated); Last update posted 2015-06-22 (Estimated); Status verified 2015-06

CONDITIONS: Female Sexual Health
MeSH Terms: interventions — Sildenafil Citrate

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (4):
- 1 (Placebo Comparator): 1 g (placebo) 0 mg sildenafil 50% external (i.e. labia minora and clitoral area) / 50% intravaginal
  Interventions: Drug: Sildenafil
- 2 (Active Comparator): 1 g 50 mg sildenafi 50% external (i.e. labia minora and clitoral area) / 50% intravaginal
  Interventions: Drug: Sildenafil
- 3 (Active Comparator): 2 g 100 mg sildenafi 50% external (i.e. labia minora and clitoral area) / 50% intravaginal
  Interventions: Drug: Sildenafil
- 4 (Active Comparator): 4 g 200 mg sildenafi 50% external (i.e. labia minora and clitoral area) / 50% intravaginal
  Interventions: Drug: Sildenafil

INTERVENTIONS:
Drug: Sildenafil

SUMMARY:
This is a Phase 1, single center, open-label, within-subject dose-escalation study evaluating the safety and pharmacokinetics of SST-6006 in healthy postmenopausal women. Three dose levels of SST-6006 and a placebo regimen will be evaluated: 1 g (0 mg of sildenafil), 1 g (50 mg of sildenafil), 2 g (100 mg of sildenafil), and 4 g (200 mg of sildenafil). Doses will be administered sequentially and will be separated by a 14-16 day washout period. All 3 dose levels and the placebo will be applied both externally and internally.

DETAILED DESCRIPTION:
Subject eligibility will be determined through Screening evaluations. Screening evaluations will include a review of inclusion and exclusion criteria, medical and Ob-Gyn history; full physical and gynecological examinations (including vulvar-vaginal examination); Pap smear; vital signs (supine); orthostatic blood pressure and heart rate; laboratory assessments (chemistry, hematology, prothrombin time, FSH and urinalysis); concomitant medication use; electrocardiogram (ECG); serology for hepatitis B surface antigen (HBsAg), hepatitis C virus (HCV) antibodies, sexually transmitted infection (syphilis, gonorrhea, chlamydia), Herpes (HSV-2) and human immunodeficiency virus (HIV) antibodies; and urine drug screen. The Screening visit will occur up to 28 days before Day 1.

For each dose level, safety from the first 2 subjects dosed will be evaluated prior to dosing the remainder of subjects at that dose level. If results indicate safety issues (defined as a known occurrence of an event of orthostatic hypotension (up to 8 hours post dose) and/or any score above 0 using the 4 point Vulvar-vaginal Irritation Scale in the first 2 subjects, an additional 2 subjects will be dosed and safety data evaluated. If no additional safety problems are found, the remaining subjects will be dosed at that level. If safety issues are found in the second 2 subjects dosed, no further dosing will occur and the prior dose level will be considered the maximum tolerated dose. In addition, any subject who experiences orthostatic hypotension at any point in the study or has a vulvar-vaginal irritation score above a 0 using the 4 point Vulvar-vaginal Irritation Scale at any dosing level will be withdrawn from the study and not proceed to the next level. An additional review of the safety data upon completion of dosing at each level will be done to determine if dose escalation is warranted. Safety decisions will be made by the Principal Investigator (PI) and the Medical Monitor based on their clinical judgment.

The first day of dosing will be considered Day 1. Subjects will be housed in the clinic for the duration of each Treatment Period to allow for collection of the PK samples up to 32 hours post-dose and the completion of all discharge procedures.

ELIGIBILITY:
Inclusion Criteria:

1. Subject must be postmenopausal (surgically induced or natural) between the ages of 35 and 65 years, inclusive, verified by 1 of the following:

   * Surgical oophorectomy, partial hysterectomy, or full hysterectomy at least 1 year prior to screening (self-report).
   * No spontaneous menses > 1 year (self-report).
2. Subject must have a serum follicle-stimulating hormone (FSH) lab result > 40mIU/mL.
3. Subject has a body mass index (BMI) from 18 to 33 kg/m², inclusive.
4. Subject has a normal electrocardiogram at baseline.
5. Subject has had a Pap smear performed within one year prior to the Screening visit and can provide documentation indicating normal test results.

   * If the subject cannot provide documentation, a Pap smear will be performed at Screening. Subjects with abnormal findings will be excluded from study participation and be referred for follow-up medical care as appropriate.
6. Subject is in good health for age, as determined by medical and Ob-Gyn history and physical and gynecological examinations.

   * As part of the gynecological exam the subject must have a pain intensity score of 0 with the cotton swab test in the lower vagina, labia majora, and labia minora when asked about pain intensity on the 0 -¬ 10 verbal rating scale when gently pressing cotton swab. Also with the cotton swab test to assess tenderness within the vulvar vestibule the score must be similarly 0 on the pain intensity score on the 0 ¬ 10 verbal rating scale when gently pressing the cotton swab at 2, 5, 7 and 10 o'clock position within the vulvar vestibule.
7. Subject is a non-smoker (no tobacco use within 6 months) and agrees not to smoke for the duration of the study up until completion of the last Treatment Period.
8. Subject is capable of understanding and complying with the protocol and agrees to sign the informed consent document.
9. Subject agrees to abstain from sexual activity (anal, oral, or vaginal) for one week after discharge for each Treatment Period to avoid potential partner exposure to the investigational product.
10. Subjects must agree to not use vaginal or vulvar lubricants, spermicides, creams or gels, foams or vaginal douche products for the duration of the study.

Exclusion Criteria:

1. Subject has any disorder or a history of any disorder that may prevent the successful completion of the study in the opinion of the PI.
2. Subject has a significant cardiovascular, hepatic, renal, respiratory, gastrointestinal, endocrine, immunologic, dermatologic, hematologic, neurologic, genitourinary, or psychiatric disease or other unstable medical condition that would contraindicate administration of study medication, interfere with study evaluation, limit study participation, or confound the interpretation of study results in the opinion of the PI.
3. Subject has a history of sexual or physical abuse.
4. Subject had an active ulcer or clinically significant bleeding disorder.
5. Subject has a history of myocardial infarction, stroke, or life-threatening arrhythmia within 6 months prior to Day 1; or any history of coronary disease causing angina; or congestive heart failure requiring medical intervention.
6. Subject has retinitis pigmentosa or sickle cell anemia or related anemias, even if the subject feels clinically well at the time of Screening. Subjects with retinitis pigmentosa will be identified by specifically asking whether they have the condition, if there are visual signs and symptoms of the condition (including questioning subjects as to whether they have difficulty seeing at night or in low light, and if they have any visual field deficits that indicate a loss of peripheral or central vision), or if there is a family history.
7. Subject has a history of orthostatic hypotension or orthostatic hypotension which is present at the Screening visit, defined as a drop in systolic blood pressure ≥ 20 mm Hg, a drop in diastolic blood pressure ≥ 10 mm Hg or experiencing lightheadedness or dizziness at 1 or 3 minutes after the change in position from supine to standing.
8. Subject has untreated hypertension.
9. Subject has type 1 or type 2 diabetes.
10. Subject has a history of cancer, other than basal cell carcinoma.
11. Subject has any surgical or medical condition that may interfere with the absorption, distribution, metabolism, or excretion of the test article in the opinion of the PI.
12. Subject has a history of drug abuse within 1 year before Day 1.
13. Subject has a history of alcoholism within 1 year before Day 1, admitted alcohol abuse, average consumption of more than 1 standard unit of alcohol per day (a standard unit equals 12 ounces of beer, 1½ ounces of 80-proof alcohol, or 6 ounces of wine).
14. Subjects who have a history of non-arteritic ischemic optic neuropathy (NAION)
15. Subject has had treatment currently or within 1 month (28 days) prior to Day 1 with any of the following: weak, moderate, and strong inhibitors and inducers of CYP3A4 and CYP2C9 enzymes (e.g., CYP3A4: ketoconazole, clarithromycin, verapamil, diltiazem, St. John's Wort / CYP2C9: fluconazole, oxandrolone, fluvastatin, and metronidazole). Any prescription, over-the-counter (OTC) medications, or herbal products taken recently or currently being taken will be screened by study personnel prior to study enrollment to confirm such drugs do not inhibit or induce the 2 enzymes listed above. If the subject takes any prescription or OTC drugs at the direction of a health care provider that are inhibitors or inducers of CYP3A4 and CYP2C9, that provider should be consulted before medications are stopped for the purposes of study participation.
16. Subject has positive findings from the urine drug screen (e.g., amphetamines, barbiturates, benzodiazepines, cannabinoids, cocaine, methadone, and opiates).
17. Subject has positive serologic findings for sexually transmitted infection (syphilis, gonorrhea, chlamydia), human immunodeficiency virus (HIV) antibodies, hepatitis B surface antigen (HBsAg), or hepatitis C virus (HCV) antibodies.
18. Subject has had an active genital herpes infection (blisters or vesicles) at any time.
19. Subject has participated in any clinical research study evaluating another investigational drug or therapy within 30 days before Day 1 (or 6 half-lives of the investigational agent, whichever is longer).
20. Subject has any abnormal findings on vulvar-vaginal examination performed during the physical and gynecological exams at Screening (e.g., genital skin breaks, irritation, dermatoses, or lesions).
21. Subject is using any intravaginal or vulvar therapies, aside from study medication
22. Subject has used any topical (e.g. vaginal) hormone replacement therapy in the past three months
23. Subject has genital piercings or plans to get genital piercings during the study period.
24. Subject has a vaginal infection including bacterial vaginosis (see Section 11.1.5) or a yeast infection. The diagnosis of yeast infections should be made by the PI based on the physical and gynecological exams; the objective is to exclude women that are symptomatic. If the woman is not complaining of symptoms but the PI observes discharge, than the vaginal wet mount test should also be performed to confirm a diagnosis of yeast infection.
25. Subject has hypersensitivity to any ingredients in the study medication or placebo (see Tables 6 and 7).

Exclusion criteria checked prior to dosing for each dosing session:

1. Subject has consumed grapefruit, grapefruit-containing products, Seville oranges, or products containing Seville oranges (e.g., orange marmalade) within 3 days before dosing in each Treatment Period. If so they should be rescheduled.
2. Subject has had an acute disease state (e.g., nausea, vomiting, fever, or diarrhea) within 7 days before Day 1.
3. Subject has any abnormal findings on vulvar-vaginal examination (e.g., genital skin breaks, irritation, dermatoses or lesions).
4. Subject must continue to not have clinical evidence of a sexually transmitted disease or a vaginal infection and must be asymptomatic of yeast and bacterial vaginosis (BV). If a subject presents with a sexually transmitted disease, vaginal, yeast or a BV infection during the study period, and the PI decides that treatment is required, the subject will be excluded for further participation in the study except if the subject has a yeast or BV infection which could be treated with Monistat one day topical treatment followed by a minimum of a two day washout for a yeast infection or 2 day oral tinidazole (i.e., Tindamax) for a BV infection. Treatment Period visits can be rescheduled to allow for treatment of yeast and BV infection.

Ages: 35 Years to 65 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 21 (Actual)
Dates: Start 2015-01; Primary Completion 2015-05 (Actual); Study Completion 2015-05 (Actual)

PRIMARY OUTCOMES:
Vaginal Irritation | 32 hours
  • Occurrence of vulvar-vaginal reactions documented on the vaginal safety questionnaire By Berger Bowman rating and AEs
Orthostatic Hypotension | 32 Hours
  Vital sign measurement
Incidence of AEs | 32 hours
  Adverse events, including occurrence of headache, orthostatic hypotension, flushing, dyspepsia, nasal congestion, urinary tract infection, abnormal vision (chromatopsia,increased sensitivity to light, blurred vision), diarrhea, dizziness, and rash

SECONDARY OUTCOMES:
Cmax, | 32 hours
  Concentration max Tmax AUC0 t AUC0-∞ Kel t1/2 Cmax Tmax AUC0 t AUC0-∞ Kel
AUC | 32 hours
  Area under curve
T 1/2 | 32 hours
  Half life

CONTACTS AND LOCATIONS:
Overall Officials: Ken Lassseter, MD, Principal Investigator — CPMI
Locations (1):
- Clinical Pharmacology of Miami, Inc., Miami, Florida, United States